CLINICAL TRIAL: NCT01575873
Title: A Randomized, Double-blind, Active-controlled Study to Evaluate the Efficacy and Safety of Denosumab Compared With Risedronate in Glucocorticoid-treated Individuals
Brief Title: Efficacy and Safety of Denosumab Compared With Risedronate in Individuals Taking Glucocorticoids
Acronym: GIOP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20101217; 2010-024393-19 (EudraCT Number)
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Steroid-induced Osteopor, Glucocorticoid-induced Ostepor
Keywords: GIOP, Glucocorticoid, osteporosis, denosumab, BMD, Bone Mineral Density
MeSH Terms: interventions — Denosumab; Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Denosumab (Experimental): Participants received 60 mg denosumab by subcutaneous injection on day 1 and at months 6, 12, and 18. Participants also received placebo to risedronate orally once a day for 24 months.
  Interventions: Drug: Denosumab; Drug: Placebo for risendronate
- Risendronate (Experimental): Participants received 5 mg risedronate orally once a day for 24 months and placebo to densumab by subcutaneous injection on day 1 and at months 6, 12, and 18.
  Interventions: Drug: Risendronate; Drug: Placebo for denosumab

INTERVENTIONS:
Drug: Denosumab — Administered by subcutaneous injection once every 6 months
  Other Names: Prolia®
  Arms: Denosumab
Drug: Placebo for risendronate — Administered orally once a day
  Arms: Denosumab
Drug: Risendronate — Administered orally once a day
  Other Names: Actonel, Atelvia
  Arms: Risendronate
Drug: Placebo for denosumab — Administered by subcutaneous injection once every 6 months
  Arms: Risendronate

SUMMARY:
This is a 2-year study to evaluate the effect of denosumab versus risedronate in adults with glucocorticoid-induced osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

Men and women 18 years of age or older who have been taking glucocorticoid treatment. Men and women who are less than 50 years of age must have had a fracture as an adult to be eligible. Men and women who are 50 years of age or older who have been taking glucocorticoids must meet protocol-specific BMD criteria.

Exclusion Criteria:

Use of agents affecting bone metabolism, use of more than one biologic agent for inflammatory disease, history of bone disease (except osteoporosis), low vitamin D level (one can enter the trial after vitamin D levels are corrected), abnormalities of blood calcium, an underactive or overactive thyroid condition that is not treated and stable, Addison's disease, any abnormality of the parathyroid glands (the glands that control blood calcium), currently pregnant or planning a pregnancy, currently breast feeding, and other criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 795 (Actual)
Dates: Start 2012-03-28 (Actual); Primary Completion 2016-06-21 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (86):
- United States (17):
  - Research Site, Birmingham, Alabama
  - Research Site, Sacramento, California
  - Research Site, Lakewood, Colorado
  - Research Site, Pembroke Pines, Florida
  - Research Site, Gainesville, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Bethesda, Maryland
  - Research Site, Cumberland, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Fargo, North Dakota
  - Research Site, Mayfield, Ohio
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Beckley, West Virginia
- Argentina (2):
  - Research Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Research Site, Buenos Aires
- Belgium (5):
  - Research Site, Brussels
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, Liège
  - Research Site, Wilrijk
- Canada (9):
  - Research Site, Vancouver, British Columbia
  - Research Site, Barrie, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Westmout, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Research Site, Barranquilla, Atlántico, Colombia
- Czechia (6):
  - Research Site, Brno
  - Research Site, Pardubice
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Praha 11 - Chodov
  - Research Site, Uherské Hradiště
- Denmark (4):
  - Research Site, Aalborg
  - Research Site, Århus C
  - Research Site, Ballerup Municipality
  - Research Site, Vejle
- France (3):
  - Research Site, Lyon Cédex 3
  - Research Site, Orléans
  - Research Site, Vandœuvre-lès-Nancy
- Germany (6):
  - Research Site, Bad Nauheim
  - Research Site, Bad Reichenhall
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Hildesheim
  - Research Site, Vogelsang-Gommern
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Gyula
  - Research Site, Szeged
  - Research Site, Szikszó
- Mexico (4):
  - Research Site, León, Guanajuato
  - Research Site, Mexico City, Mexico City
  - Research Site, Morelia, Michoacán
  - Research Site, San Luis Potosí City, San Luis Potosí
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Helmond
  - Research Site, Utrecht
- Poland (8):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Stalowa Wola
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (5):
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- South Korea (5):
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Gwangju
  - Research Site, Jinju
  - Research Site, Seoul
- Spain (3):
  - Research Site, Barcelona, Catalonia
  - Research Site, Valencia, Valencia
  - Research Site, Madrid

REFERENCES:
- [Background] Saag KG, Wagman RB, Geusens P, Adachi JD, Messina OD, Emkey R, Chapurlat R, Wang A, Pannacciulli N, Lems WF. Denosumab versus risedronate in glucocorticoid-induced osteoporosis: a multicentre, randomised, double-blind, active-controlled, double-dummy, non-inferiority study. Lancet Diabetes Endocrinol. 2018 Jun;6(6):445-454. doi: 10.1016/S2213-8587(18)30075-5. Epub 2018 Apr 6. PMID 29631782
- [Derived] Saag KG, Pannacciulli N, Geusens P, Adachi JD, Messina OD, Morales-Torres J, Emkey R, Butler PW, Yin X, Lems WF. Denosumab Versus Risedronate in Glucocorticoid-Induced Osteoporosis: Final Results of a Twenty-Four-Month Randomized, Double-Blind, Double-Dummy Trial. Arthritis Rheumatol. 2019 Jul;71(7):1174-1184. doi: 10.1002/art.40874. Epub 2019 May 25. PMID 30816640
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 79 centers in Europe, North America, Latin America, and Korea from 28 March 2012 to 30 June 2015.
  Participants who had been taking glucocorticoids for at least 3 months were classed as glucocorticoid continuing; those who were taking glucocorticoids for less than 3 months were classed as glucocorticoid initiating.
Pre-assignment Details: Eligible patients were randomly assigned in a 1:1 ratio to receive 60 mg denosumab every 6 months or 5 mg oral risedronate daily for 24 months within each subpopulation. Randomization was stratified by sex within each subpopulation.
Groups:
- Risedronate: Glucocorticoid-initiating; Risedronate: Glucocorticoid-continuing: Participants received 5 mg risedronate orally once a day for 24 months and placebo to densumab by subcutaneous injection on day 1 and at months 6, 12, and 18.
- Denosumab: Glucocorticoid-initiating; Denosumab: Glucocorticoid-continuing: Participants received 60 mg denosumab by subcutaneous injection on day 1 and at months 6, 12, and 18. Participants also received placebo to risedronate orally once a day for 24 months.
Period: Overall Study
Arm/Group | Risedronate: Glucocorticoid-initiating | Denosumab: Glucocorticoid-initiating | Risedronate: Glucocorticoid-continuing | Denosumab: Glucocorticoid-continuing
Started | 145 | 145 | 252 | 253
Received Study Drug | 140 (Participants who received oral risedronate) | 142 (Participants who received subcutaneous denosumab) | 246 (Participants who received oral risedronate) | 251 (Participants who received subcutaneous denosumab)
Completed | 117 | 109 | 178 | 186
Not Completed | 28 | 36 | 74 | 67
Not completed — Withdrawal by Subject | 15 | 20 | 34 | 34
Not completed — Adverse Event | 7 | 7 | 9 | 12
Not completed — Lost to Follow-up | 1 | 3 | 13 | 5
Not completed — Death | 3 | 2 | 8 | 9
Not completed — Noncompliance | 1 | 2 | 4 | 3
Not completed — Administrative decision | 1 | 1 | 1 | 0
Not completed — Protocol deviation | 0 | 1 | 0 | 1
Not completed — Requirement for Alternative Therapy | 0 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Risedronate: Glucocorticoid-initiating | Denosumab: Glucocorticoid-initiating | Risedronate: Glucocorticoid-continuing | Denosumab: Glucocorticoid-continuing | Total
Number analyzed (Participants) | 145 | 145 | 252 | 253 | 795
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (10.0) | 67.5 (10.1) | 61.3 (11.1) | 61.5 (11.6) | 63.1 (11.1)
Age, Customized [Count of Participants; unit: Participants]
  < 50 years | 5 | 2 | 26 | 33 | 66
  50 - 64 years | 75 | 55 | 130 | 114 | 374
  65 - 74 years | 38 | 50 | 62 | 73 | 223
  ≥ 75 years | 27 | 38 | 34 | 33 | 132
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 93 | 185 | 185 | 556
  Male | 52 | 52 | 67 | 68 | 239
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 20 | 54 | 43 | 135
  Not Hispanic or Latino | 127 | 125 | 198 | 210 | 660
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 123 | 122 | 223 | 230 | 698
  Other | 11 | 12 | 11 | 13 | 47
  Asian | 9 | 9 | 12 | 6 | 36
  Black or African American | 2 | 2 | 4 | 4 | 12
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Multiple | 0 | 0 | 1 | 0 | 1
Menopausal Status [Count of Participants; unit: Participants] — Population: Females only
  Participants
    number analyzed (Participants) | 93 | 93 | 185 | 185 | 556
    Premenopause | 7 | 10 | 25 | 24 | 66
    Postmenopause | 83 | 82 | 157 | 159 | 481
    Unknown | 3 | 1 | 3 | 2 | 9
Lumbar Spine Bone Mineral Density (BMD) T-score [Mean (Standard Deviation); unit: T-score] — The T-score is the bone mineral density (BMD) at the site when compared to that of a healthy thirty-year-old. Normal is a T-score of -1.0 or higher; Osteopenia is defined as between -1.0 and -2.5; Osteoporosis is defined as -2.5 or lower, meaning a bone density that is two and a half standard deviations below the mean of a thirty-year-old man/woman. Population: Participants with observed values
  T-score
    Glucocorticoid-initiating Subpopulation: number analyzed (Participants) | 143 | 144 | 0 | 0 | 287
    Glucocorticoid-initiating Subpopulation | -1.06 (1.57) | -0.92 (1.86) |  |  | -0.99 (1.72)
    Glucocorticoid-continuing Subpopulation: number analyzed (Participants) | 0 | 0 | 252 | 249 | 501
    Glucocorticoid-continuing Subpopulation |  |  | -1.96 (1.38) | -1.92 (1.38) | -1.94 (1.38)
Total Hip BMD T-score [Mean (Standard Deviation); unit: T-score] — The T-score is the bone mineral density (BMD) at the site when compared to that of a healthy thirty-year-old. Normal is a T-score of -1.0 or higher; Osteopenia is defined as between -1.0 and -2.5; Osteoporosis is defined as -2.5 or lower, meaning a bone density that is two and a half standard deviations below the mean of a thirty-year-old man/woman. Population: participants with observed vaues
  T-score
    Glucocorticoid-initiating Subpopulation: number analyzed (Participants) | 142 | 142 | 0 | 0 | 284
    Glucocorticoid-initiating Subpopulation | -0.98 (1.07) | -1.14 (1.00) |  |  | -1.06 (1.04)
    Glucocorticoid-continuing Subpopulation: number analyzed (Participants) | 0 | 0 | 250 | 249 | 499
    Glucocorticoid-continuing Subpopulation |  |  | -1.56 (0.96) | -1.66 (0.96) | -1.61 (0.96)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density at Month 12 (Non-inferiority Analysis)
Description: Bone mineral density at the lumbar spine was measured by dual-energy x-ray absorptiometry (DXA).
Time Frame: Baseline and month 12
Population: Randomized participants with a baseline and month 12 measurement for the lumbar spine BMD.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Risedronate: Glucocorticoid-initiating | Denosumab: Glucocorticoid-initiating | Risedronate: Glucocorticoid-continuing | Denosumab: Glucocorticoid-continuing
Number analyzed (Participants) | 126 | 119 | 211 | 209
percent change | 0.8 [0.2 to 1.5] | 3.8 [3.1 to 4.5] | 2.3 [1.7 to 2.9] | 4.4 [3.8 to 5.0]
Statistical Analysis 1: Comparison: Risedronate: Glucocorticoid-initiating vs Denosumab: Glucocorticoid-initiating; Analyses of the primary and secondary endpoints were performed independently within the glucocorticoid-continuing and glucocorticoid-initiating subpopulations. A fixed-sequence testing procedure was used to control the experiment-wise type 1 error rate at a two-sided 5% significance level within each subpopulation. The glucocorticoid-initiating subpopulation was analyzed using an ANCOVA model adjusting for treatment, baseline BMD, sex, machine type, and baseline BMD-by-machine type interaction; Test type: Non-Inferiority — Non-inferiority was shown if the lower bound of the two-sided 95% CI for the difference between the least-squares means (denosumab minus risedronate) was higher than the prespecified non-inferiority margin of -1.1 percentage points for the glucocorticoid-initiating subpopulation; p < 0.001, ANCOVA — One-sided p-value based on the prespecified noninferiority margin for lumbar spine of -1.1%; LS Mean Difference = 2.9, 95% CI 2-sided [2.0 to 3.9] — Least Squares (LS) Mean Difference = Denosumab - Risedronate
Statistical Analysis 2: Comparison: Risedronate: Glucocorticoid-continuing vs Denosumab: Glucocorticoid-continuing; Analyses of the primary and secondary endpoints were performed independently within each subpopulation using a fixed-sequence testing procedure to control the experiment-wise type 1 error rate at a two-sided 5% significance level. The glucocorticoid-continuing subpopulation was analyzed using an ANCOVA model adjusted for treatment, baseline BMD, sex, machine type, baseline BMD-by-machine type interaction, and duration of prior glucocorticoid use (< 12 months vs ≥ 12 months); Test type: Non-Inferiority — Non-inferiority was shown if the lower bound of the two-sided 95% CI for the difference between the least-squares means (denosumab minus risedronate) was higher than the prespecified non-inferiority margin of -0.7 percentage points for the glucocorticoid-continuing subpopulation; p < 0.001, ANCOVA — One-sided p-value based on the prespecified noninferiority margins for lumbar spine of -0.7%; LS Mean Difference = 2.2, 95% CI 2-sided [1.4 to 3.0] — LS Mean Difference = Denosumab - Risedronate

2. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density at Month 12 (Superiority Analysis)
Description: Bone mineral density at the lumbar spine was measured by dual-energy x-ray absorptiometry (DXA).
Time Frame: Baseline and month 12
Population: Randomized participants with a baseline and month 12 measurement for the lumbar spine BMD.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Risedronate: Glucocorticoid-initiating | Denosumab: Glucocorticoid-initiating | Risedronate: Glucocorticoid-continuing | Denosumab: Glucocorticoid-continuing
Number analyzed (Participants) | 126 | 119 | 211 | 209
percent change | 0.8 [0.2 to 1.5] | 3.8 [3.1 to 4.5] | 2.3 [1.7 to 2.9] | 4.4 [3.8 to 5.0]
Statistical Analysis 1: Comparison: Risedronate: Glucocorticoid-initiating vs Denosumab: Glucocorticoid-initiating; Analyses of the primary and secondary endpoints were performed independently within each subpopulation using a fixed-sequence testing procedure to control the experiment-wise type 1 error rate at a two-sided 5% significance level. The glucocorticoid-initiating subpopulation was analyzed using an ANCOVA model adjusting for treatment, baseline BMD value, sex, machine type, and baseline BMD value-by-machine type interaction; Test type: Superiority; p < 0.001, ANCOVA — 2-sided p-value corresponding to the 2-sided 95% confidence interval; LS Mean Difference = 2.9, 95% CI 2-sided [2.0 to 3.9] — LS Mean Difference = Denosumab - Risedronate
Statistical Analysis 2: Comparison: Risedronate: Glucocorticoid-continuing vs Denosumab: Glucocorticoid-continuing; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA — 2-sided p-value corresponding to the 2-sided 95% confidence interval; LS Mean Difference = 2.2, 95% CI 2-sided [1.4 to 3.0] — LS Mean Difference = Denosumab - Risedronate

3. Secondary Outcome: Percent Change From Baseline in Total Hip Bone Mineral Density at Month 12
Description: Bone mineral density at the total hip was measured by dual-energy x-ray absorptiometry (DXA).
Time Frame: Baseline and month 12
Population: Randomized participants with a baseline and month 12 measurement for the total hip BMD.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Risedronate: Glucocorticoid-initiating | Denosumab: Glucocorticoid-initiating | Risedronate: Glucocorticoid-continuing | Denosumab: Glucocorticoid-continuing
Number analyzed (Participants) | 128 | 119 | 215 | 217
percent change | 0.2 [-0.2 to 0.7] | 1.7 [1.2 to 2.2] | 0.6 [0.2 to 1.0] | 2.1 [1.7 to 2.5]
Statistical Analysis 1: Comparison: Risedronate: Glucocorticoid-initiating vs Denosumab: Glucocorticoid-initiating; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA — 2-sided p-value corresponding to the 2-sided 95% confidence interval; LS Mean Difference = 1.5, 95% CI 2-sided [0.8 to 2.1] — LS Mean Difference = Denosumab - Risedronate
Statistical Analysis 2: Comparison: Risedronate: Glucocorticoid-continuing vs Denosumab: Glucocorticoid-continuing; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA — 2-sided p-value corresponding to the 2-sided 95% confidence interval; LS Mean Difference = 1.5, 95% CI 2-sided [1.0 to 2.1] — LS Mean Difference = Denosumab - Risedronate

4. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density at Month 24
Description: Bone mineral density at the lumbar spine was measured by dual-energy x-ray absorptiometry (DXA).
Time Frame: Baseline and month 24
Population: Randomized participants with a baseline and month 24 measurement for the lumbar spine BMD.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Risedronate: Glucocorticoid-initiating | Denosumab: Glucocorticoid-initiating | Risedronate: Glucocorticoid-continuing | Denosumab: Glucocorticoid-continuing
Number analyzed (Participants) | 113 | 107 | 174 | 183
percent change | 1.7 [0.8 to 2.7] | 6.2 [5.3 to 7.2] | 3.2 [2.3 to 4.1] | 6.4 [5.5 to 7.2]
Statistical Analysis 1: Comparison: Risedronate: Glucocorticoid-initiating vs Denosumab: Glucocorticoid-initiating; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA — 2-sided p-value corresponding to the 2-sided 95% confidence interval; LS Mean Difference = 4.5, 95% CI 2-sided [3.2 to 5.8] — LS Mean Difference = Denosumab - Risedronate
Statistical Analysis 2: Comparison: Risedronate: Glucocorticoid-continuing vs Denosumab: Glucocorticoid-continuing; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA — 2-sided p-value corresponding to the 2-sided 95% confidence interval; LS Mean Difference = 3.2, 95% CI 2-sided [2.0 to 4.3] — LS Mean Difference = Denosumab - Risedronate

5. Secondary Outcome: Percent Change From Baseline in Total Hip Bone Mineral Density at Month 24
Description: Bone mineral density at the total hip was measured by dual-energy x-ray absorptiometry (DXA).
Time Frame: Baseline and month 24
Population: Randomized participants with a baseline and month 24 measurement for the total hip BMD.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Risedronate: Glucocorticoid-initiating | Denosumab: Glucocorticoid-initiating | Risedronate: Glucocorticoid-continuing | Denosumab: Glucocorticoid-continuing
Number analyzed (Participants) | 111 | 104 | 176 | 181
percent change | -0.0 [-0.6 to 0.6] | 3.1 [2.4 to 3.7] | 0.5 [-0.1 to 1.0] | 2.9 [2.4 to 3.5]
Statistical Analysis 1: Comparison: Risedronate: Glucocorticoid-initiating vs Denosumab: Glucocorticoid-initiating; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA — 2-sided p-value corresponding to the 2-sided 95% confidence interval; LS Mean Difference = 3.1, 95% CI 2-sided [2.2 to 3.9] — LS Mean Difference = Denosumab - Risedronate
Statistical Analysis 2: Comparison: Risedronate: Glucocorticoid-continuing vs Denosumab: Glucocorticoid-continuing; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA — 2-sided p-value corresponding to the 2-sided 95% confidence interval; LS Mean Difference = 2.5, 95% CI 2-sided [1.7 to 3.2] — LS Mean Difference = Denosumab - Risedronate

ADVERSE EVENTS:
Time Frame: 24 months.
Description: One participant was randomized to risedronate but received denosumab in error; this participant was included in the denosumab group for safety analyses.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Risedronate: Participants received 5 mg risedronate orally once a day for 24 months and placebo to densumab by subcutaneous injection on day 1 and at months 6, 12, and 18.
Arm/Group | Risedronate | Denosumab
All-Cause Mortality (participants affected / at risk) | 9/385 | 13/394
Serious Adverse Events (participants affected / at risk) | 98/385 | 92/394
Other Adverse Events (participants affected / at risk) | 76/385 | 77/394
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Risedronate (N=385) | Denosumab (N=394)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Aortic valve sclerosis (Cardiac disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 3
Cardiac failure acute (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 2 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Mitral valve disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 2
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Congenital megaureter (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 2 | 1
Glaucoma (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Colitis ulcerative (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Lumbar hernia (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 2 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Death (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Eosinophilic granulomatosis with polyangiitis (Immune system disorders) | 1 | 0
Food allergy (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium colitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 2
Erysipelas (Infections and infestations) | 1 | 2
Escherichia sepsis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Haemorrhagic fever (Infections and infestations) | 0 | 1
Helicobacter gastritis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1
Lymph node tuberculosis (Infections and infestations) | 0 | 1
Lymphangitis (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 8 | 7
Pneumonia bacterial (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 2 | 0
Septic shock (Infections and infestations) | 1 | 0
Serratia infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Wound infection bacterial (Infections and infestations) | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 3
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Ketosis (Metabolism and nutrition disorders) | 1 | 0
Periarthritis calcarea (Metabolism and nutrition disorders) | 1 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Exposed bone in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Ataxia (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 3
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0
Paresis (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 2
Seizure (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 1 | 0
Behaviour disorder due to a general medical condition (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Lupus nephritis (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Cervix haematoma uterine (Reproductive system and breast disorders) | 0 | 1
Cystocele (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Cataract operation (Surgical and medical procedures) | 1 | 0
Colectomy (Surgical and medical procedures) | 1 | 0
Ileostomy (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 2 | 1
Lung neoplasm surgery (Surgical and medical procedures) | 1 | 0
Lymphadenectomy (Surgical and medical procedures) | 0 | 1
Sigmoidectomy (Surgical and medical procedures) | 0 | 1
Spinal decompression (Surgical and medical procedures) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Haemodynamic instability (Vascular disorders) | 1 | 0
Temporal arteritis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Risedronate (N=385) | Denosumab (N=394)
Viral upper respiratory tract infection (Infections and infestations) | 19 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 24
Hypertension (Vascular disorders) | 15 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.